CLINICAL TRIAL: NCT02919293
Title: Immunogenicity and Safety of Adjuvant and Adjuvant-Free Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine in Infants 2 to 5 Months of Age
Brief Title: Immunogenicity and Safety of Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine in Infants 2 to 5 Months of Age
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Collaborators: Guangdong Center for Disease Prevention and Control (Other Government); Guizhou Center for Disease Control and Prevention (Other); National Institutes for Food and Drug Control, China (Other); Air Force Military Medical University, China (Other); Simoon Record Pharma Information Consulting Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 085201602
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant-Free MenAC-Hib Conjugate Vaccine Group (Experimental): Participants randomized to receive adjuvant-free MenAC-Hib conjugate vaccine.
  Interventions: Biological: Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine (adjuvant-free)
- Adjuvant MenAC-Hib Conjugate Vaccine Group (Active Comparator): Participants randomized to receive adjuvant MenAC-Hib conjugate vaccine.
  Interventions: Biological: Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine(adjuvant)

INTERVENTIONS:
Biological: Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine (adjuvant-free) — 30μg /dose, Intramuscular
  Other Names: HibACon; MenAC-Hib
  Arms: Adjuvant-Free MenAC-Hib Conjugate Vaccine Group
Biological: Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine(adjuvant) — 0.5ml /dose, Intramuscular
  Other Names: HibACon; MenAC-Hib
  Arms: Adjuvant MenAC-Hib Conjugate Vaccine Group

SUMMARY:
To evaluate Immunogenicity and Safety of Adjuvant and Adjuvant-Free Meningococcal Groups A and C and Haemophilus b Conjugate Vaccine in Infants 2 to 5 Months of Age.

Primary objective:

* To demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C and Haemophilus influenzae type b following the administration of adjuvant-free MenAC-Hib conjugate vaccine compared to those observed following the administration of adjuvant MenAC-Hib conjugate vaccine.
* To describe the safety profile of adjuvant-free MenAC-Hib conjugate vaccine compared to that of adjuvant MenAC-Hib conjugate vaccine.

Secondary objective:

•To compare the antibody level of meningococcal serogroups A, C and Haemophilus influenzae type b following the administration of adjuvant-free MenAC-Hib conjugate vaccine to those observed following the administration of adjuvant MenAC-Hib conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Health infants aged 2 to 5 months.
* Legal guardian has signed written informed consent.
* Guardian may finish the whole visit in the judgment of investigator.
* 2-5 months health infants who haven't immuned with any Meningococcal A and C Conjugate Vaccine or Haemophilus b Conjugate Vaccine.
* Subject who did't vaccinated with any live vaccine within 14 days or inactivated vaccine within 10 days before vaccination.

Exclusion Criteria:

* Fever, body temperature ≥37.1℃.
* History of severe allergic reaction that needs medical intervention including throat swelling, dyspnea, hypotension or shock; History of allergic reaction to vaccine or to any of the vaccine components especially to tetanus toxoid or history of other severe adverse reaction to vaccine.
* Clear diagnosis of thrombocytopenia or history of other coagulation disorders that may cause contraindications of intramuscular injection.
* Subject with history of abnormal labor, asphyxia rescue history,congenital malformations,eccyliosis or severe chronic disease.
* Severe cardiovascular or liver and kidney disease, active tuberculosis and HIV infection.
* Subject with encephalopathy, uncontrolled epilepsy and other progressive nervous system disease.
* Subject suffer from acute disease, severe chronic disease, acute episode of chronic disease and febrile illness (temperature ≥ 38°C) within 3 days.
* Any condition that, in the judgment of investigator, subject is not suitable for participation in this clinical trial.

Ages: 2 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with seroresponse to meningococcal serogroups A,C and Haemophilus b post-vaccination with 3 doses of MenAC-Hib conjugate vaccine | Day 30 post-vaccination
Occurrence of adverse events during a 30 day follow-up period after each vaccination | 30 day after each vaccination

SECONDARY OUTCOMES:
Occurrence of severe adverse events within six months post-vaccination | six months post-vaccination
Geometric mean titer （GMT）of antibodies against meningococcal serogroups A, C and Haemophilus b post-vaccination with 3 doses of MenAC-Hib conjugate vaccine | Day 30 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Gaozhou Center for Disease Control and Prevention, Gaozhou, Guangdong, China